CLINICAL TRIAL: NCT04954560
Title: Losartan and Eprosartan Induce a Similar Effect on Oral Fructose-induced Rise in Serum Uric Acid Concentration in Patients With Metabolic Syndrome
Brief Title: Effect of Losartan or Eprosartan on Fructose Hyperuricemia
Acronym: metabolic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Lodz (Other)
Responsible Party: Principal Investigator, Michal Nowicki, Profesor, Medical University of Lodz
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RNN/185/07/KE
Record Dates: First submitted 2021-06-03; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-06

CONDITIONS: Uric Acid Concentration, Serum, Quantitative Trait Locus 7
Keywords: sartan; fructose; metabolic syndrome; uric acid
MeSH Terms: conditions — Metabolic Syndrome | interventions — Losartan; eprosartan

STUDY DESIGN:
Intervention Model Description: The study was designed as a randomized, crossover, head-to-head comparative study. Randomization was carried out using MS Excel random number generator. After qualification each patient was randomly assigned to receive either losartan (Lorista, KRKA, Slovenia) or eprosartan (Teveten, Solvay Pharmaceuticals, Austral-ia). The patients were taking all other previously prescribed drugs in unmodified dos-es during the whole course of the study. Each study drug was given in a random or-der as a single morning dose (50 mg of losartan or 600 mg of eprosartan) for two periods each lasting 3 months separated by 2-week wash-out time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- losartan (Active Comparator): Each study drug was given in a random order as a single morning dose (50 mg of losartan or 600 mg of eprosartan) for two periods each lasting 3 months separated by 2-week wash-out time.
  Interventions: Drug: losartan and eprosartan
- eprosartan (Active Comparator): Each study drug was given in a random order as a single morning dose (50 mg of losartan or 600 mg of eprosartan) for two periods each lasting 3 months separated by 2-week wash-out time.
  Interventions: Drug: losartan and eprosartan

INTERVENTIONS:
Drug: losartan and eprosartan — . Each study drug was given in a random order as a single morning dose (50 mg of losartan or 600 mg of eprosartan) for two periods each lasting 3 months separated by 2-week wash-out time.
  Other Names: Lorista; Teveten

SUMMARY:
Hyperuricemia is seen in about 20% of adults in the general population, Chronic hyperuricemia, frequently manifesting as the gout, is a well-known risk factor of joint damage but has been also linked to a variety of other pathologies mostly affecting the cardiovascular system. The close relation between high uric acid concentration and increased risk of cardiovascular disease has been reported for more than a century. Furthermore, many studies reported a strong association between hyperuricemia, arterial hypertension, obesity and cardiovascular diseases even in an absence of typical clinical manifestations of gout.

Several studies showed that the prevalence of hyperuricemia in patients with hypertension is much higher than in the general population and may worsen after the onset of antihypertensive treatment. That may indicate that hyperuricemia may be also caused by antihypertensive drugs. In contrast to diuretics and nonselective beta blockers the agents that block the renin-angiotensin-aldosterone system have had a neutral effect on serum uric acid. Several clinical studies showed that losartan in contrast to other AT1-receptor agonists, may have specific uricosuric properties and thereby can lower uric acid concentration. It has been speculated that uricosuric effect could make losartan particularly useful for the treatment of arterial hypertension associated with hyperuricemia and metabolic syndrome.

The uricosuric effect of losartan is most likely due to overlapping two different mechanisms regulating the excretion of uric acid. Losartan may increase uric acid tubular secretion in the same way as other inhibitors of the renin-angiotensin-aldosterone system, but in addition it may specifically inhibit post-secretory resorption of uric acid in the proximal tubule. The effect may be due to a specific structure of the losartan molecule. The urateanion transporter is a monoammonium selective transporter, and the losartan molecule is mainly a monoanion at normal pH range (as opposed to dianion e.g. eprosartan) and therefore is a good substrate for the exchanger. However, this concept remains speculative since, e.g. irbesartan which is also a monoanion has no consistent uricosuric effect.

Fructose, in contrast to other carbohydrates causes an increase of serum uric acid concentration, which may facilitate the development of the metabolic syndrome.

DETAILED DESCRIPTION:
The study group included 16 patients (15F, 1M, mean age 64.5 ± 9.8 years). The patients selected for the study fulfilled the AHA/NHLBI 2005 criteria of the meta-bolic syndrome [30] and ESC/ESH criteria of arterial hypertension. The exclusion cri-teria included an antihypertensive therapy with the renin-angiotensin-aldosterone axis blocking agent used anytime during last 3 months, current or past therapy with SGLT2 inhibitor, GLP-1 agonist or DPP4-inhibitor, suspected or confirmed secondary form of hypertension, estimated glomerular filtration rate <60 ml/min/1.73 m2, chron-ic liver disease, acute infection, psychiatric disorders, mean serum potassium con-centration at last three measurements <4.0 mmol/l, or aspartate aminotransferase or alanine aminotransferase or creatinine kinase > x1.5 upper range limit were excluded. Seven patients had diabetes mellitus of which 4 were treated with insulin. Twelve pa-tients were receiving metformin. Waist circumference was measured on the initial visit. Plasma lipids and blood glucose were measured in a fasting state during the study.

The study was designed as a randomized, crossover, head-to-head comparative study. Randomization was carried out using MS Excel random number generator. After qualification each patient was randomly assigned to receive either losartan (Lorista, KRKA, Slovenia) or eprosartan (Teveten, Solvay Pharmaceuticals, Austral-ia). The patients were taking all other previously prescribed drugs in unmodified dos-es during the whole course of the study. Each study drug was given in a random or-der as a single morning dose (50 mg of losartan or 600 mg of eprosartan) for two periods each lasting 3 months separated by 2-week wash-out time.

Oral fructose tolerance with the administration of 75 g of fructose was con-ducted 3 times during the study in each patient, i.e. at baseline and after each of the treatment periods. Before the commencement of OFTT, the patients collected the urine for 2 hours for assessment of the urinary excretion of uric acid and creatinine. Other baseline measurements included blood pressure, serum concentration of glu-cose, uric acid, creatinine and plasma lipids (total, HDL- and, LDL-cholesterol and triglycerides). Subsequent blood samples were taken three times during each OFTT, i.e. after 30, 60 and 120 minutes from its start to determine serum uric acid concen-tration. In addition, peripheral blood pressure was measured before the collection of each blood sample. After 120 minutes blood was also taken to assess plasma lipids. The second timed 2-hour urine collection was obtained during OFTT. The same pro-cedures were repeated after each treatment period. The patients took all their pre-scribed medication including the study drug in the morning 120 minutes before the beginning of OFTT Routine automated laboratory tests were used to assess blood and urine pa-rameters. Blood pressure was taken in a sitting position with the aneroid sphygmo-manometer. Blood pressure was measured both at baseline and after 3-month ther-apy with each study drug. The mean from four measurements obtained between 0 and 120 minutes OFTT was taken for the analysis. Blood pressure was measured by a designated single member of the staff. Mean blood pressure (MAP) was calculated for all measurements as diastolic BP + 1/3 of pulse pressure (systolic BP - diastolic BP).

The results are expressed as mean ± SD or median with interquartile range depending on each variable distribution. 95% confidence intervals were calculated for the changes of the parameters caused by the treatment. Statistical significance was defined at p<0.05. The within-group comparisons were analyzed using one-way ANOVA and t-test for normally distributed variables or alternatively with non-parametric Wilcoxon test. The normality of the variable distribution was checked with Shapiro-Wilk test. The Pearson or Spearman correlation coefficient was used to as-sess the relations between variables depending on their distribution. Area under the curve (AUC) of serum uric acid during oral fructose tolerance test was calculated using the trapezoidal rule.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years old
* Fulfillment of three or more of the AHA / NHLBI 2005 assessment criteria for the metabolic syndrome:
* abdominal obesity (i.e. handling in women ≥88 cm) male ≥ 102 cm
* concentration of triglycerides in the form ≥150 mg / dl
* concentration of HDL fraction (men <40 mg / dL, women <50 mg / dL)
* blood pressure ≥ 130/85 mmHg
* Correction of fasting glucose ≥100 mg / dL)
* Written and informed consent to participate in the case of

Exclusion Criteria:

* Congenital defects in fructose metabolism (hereditary fructose intolerance and idiopathic fructosuria)
* Mental illness, dementia
* Insufficient cooperation with the patient, non-compliance with doctor's recommendations
* Pregnancy
* Bilateral renal artery stenosis or stenosis to a solitary kidney and other contraindications for angiotensin receptor antagonists
* Chronic use of uricosuric drugs, xanthine oxidase inhibitors and AT1 receptor inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2010-01-01 (Actual); Study Completion 2010-01-01 (Actual)

PRIMARY OUTCOMES:
serum uric acid after losartan | 3 months
  serum uric acid after losartan therapy
serum uric acid after eprosartan | 3 months
  serum uric acid after eprosartan therapy
urine uric acid after losartan | 3 months
  urine uric acid after losartan therapy
urine uric acid after eprosartan | 3 months
  urine uric acid after eprosartan therapy

CONTACTS AND LOCATIONS:
Overall Officials: Ireneusz Staroń, Study Chair — Medical University of Lodz

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Masajtis-Zagajewska A, Majer J, Nowicki M. Losartan and Eprosartan Induce a Similar Effect on the Acute Rise in Serum Uric Acid Concentration after an Oral Fructose Load in Patients with Metabolic Syndrome. J Renin Angiotensin Aldosterone Syst. 2021 Aug 25;2021:2214978. doi: 10.1155/2021/2214978. eCollection 2021. PMID 34527078